CLINICAL TRIAL: NCT07022522
Title: Frequency-dependent Modulation of Inhibitory Control Via Subthalamic Nucleus Subregional Stimulation in Parkinson's Disease
Brief Title: Impact of Frequency-specific Subthalamic Nucleus Subregion Stimulation on Inhibitory Control in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Jianguo Zhang, Director of Department of Functional Neurosurgery, Beijing Tiantan Hospital, Capital Medical University, Beijing, China, Beijing Tiantan Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KY2024-163-02
Record Dates: First submitted 2025-05-29; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease; Deep Brain Stimulation
Keywords: Deep Brain Stimulation; Cognition; Subthalamic Nucleus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- No stimulation (Sham Comparator)
  Interventions: Device: No stimulation
- 5Hz stimulation on the STN motor subregion (Experimental): In this experimental arm, Parkinson's disease patients will undergo deep brain stimulation targeting the motor subregion of the subthalamic nucleus at a low frequency of 5Hz, with the primary objective of evaluating its specific effects on cognitive and behavioral outcomes such as inhibitory control and reaction time. The intervention involves precise postoperative programming of DBS electrodes localized to the motor subregion using neuroimaging verification.
  Interventions: Device: 5Hz stimulation on the STN motor subregion
- 5Hz stimulation on the STN associative subregion (Experimental): In this experimental arm, Parkinson's disease patients will undergo deep brain stimulation targeting the associative subregion of the subthalamic nucleus at a low frequency of 5Hz, with the primary objective of evaluating its specific effects on cognitive and behavioral outcomes such as inhibitory control and reaction time. The intervention involves precise postoperative programming of DBS electrodes localized to the associative subregion using neuroimaging verification.
  Interventions: Device: 5Hz stimulation on the STN associative subregion
- 130Hz stimulation on the STN motor subregion (Experimental): In this experimental arm, Parkinson's disease patients will undergo deep brain stimulation targeting the motor subregion of the subthalamic nucleus at a high frequency of 130Hz, with the primary objective of evaluating its specific effects on cognitive and behavioral outcomes such as inhibitory control and reaction time. The intervention involves precise postoperative programming of DBS electrodes localized to the motor subregion using neuroimaging verification.
  Interventions: Device: 130Hz stimulation on the STN motor subregion
- 130Hz stimulation on the STN associative subregion (Experimental): In this experimental arm, Parkinson's disease patients will undergo deep brain stimulation targeting the associative subregion of the subthalamic nucleus at a high frequency of 130Hz, with the primary objective of evaluating its specific effects on cognitive and behavioral outcomes such as inhibitory control and reaction time. The intervention involves precise postoperative programming of DBS electrodes localized to the associative subregion using neuroimaging verification.
  Interventions: Device: 130Hz stimulation on the STN associative subregion

INTERVENTIONS:
Device: 5Hz stimulation on the STN motor subregion — In this experimental arm, Parkinson's disease patients will undergo deep brain stimulation targeting the motor subregion of the subthalamic nucleus at a low frequency of 5Hz, with the primary objective of evaluating its specific effects on cognitive and behavioral outcomes such as inhibitory control and reaction time. The intervention involves precise postoperative programming of DBS electrodes localized to the motor subregion using neuroimaging verification.
  Arms: 5Hz stimulation on the STN motor subregion
Device: 5Hz stimulation on the STN associative subregion — In this experimental arm, Parkinson's disease patients will undergo deep brain stimulation targeting the associative subregion of the subthalamic nucleus at a low frequency of 5Hz, with the primary objective of evaluating its specific effects on cognitive and behavioral outcomes such as inhibitory control and reaction time. The intervention involves precise postoperative programming of DBS electrodes localized to the associative subregion using neuroimaging verification.
  Arms: 5Hz stimulation on the STN associative subregion
Device: 130Hz stimulation on the STN motor subregion — In this experimental arm, Parkinson's disease patients will undergo deep brain stimulation targeting the motor subregion of the subthalamic nucleus at a high frequency of 130Hz, with the primary objective of evaluating its specific effects on cognitive and behavioral outcomes such as inhibitory control and reaction time. The intervention involves precise postoperative programming of DBS electrodes localized to the motor subregion using neuroimaging verification.
  Arms: 130Hz stimulation on the STN motor subregion
Device: 130Hz stimulation on the STN associative subregion — In this experimental arm, Parkinson's disease patients will undergo deep brain stimulation targeting the associative subregion of the subthalamic nucleus at a high frequency of 130Hz, with the primary objective of evaluating its specific effects on cognitive and behavioral outcomes such as inhibitory control and reaction time. The intervention involves precise postoperative programming of DBS electrodes localized to the associative subregion using neuroimaging verification.
  Arms: 130Hz stimulation on the STN associative subregion
Device: No stimulation — In this control arm, Parkinson's disease patients will not receive active deep brain stimulation, with the DBS system maintained in an "off" state throughout the testing period.
  Arms: No stimulation

SUMMARY:
The core symptoms of Parkinson's disease (PD) include both motor and non-motor symptoms. Cognitive impairment is one of the most common non-motor symptoms in PD patients, with approximately 30% of patients exhibiting cognitive dysfunction at diagnosis and up to 80% eventually progressing to dementia. Among these, impairment of inhibitory control is the most detrimental cognitive dysfunction, as patients with compromised inhibitory control have difficulty suppressing impulsive behaviors and maintaining attention, which severely reduces their quality of life.

The subthalamic nucleus (STN) plays an important role in the development and progression of PD. Along its longitudinal axis from posterior to anterior, it can be divided into three subregions: motor, associative, and limbic. The motor subregion receives extensive projections from the motor cortex and serves as a core node in the PD motor network, participating in the coordination and control of motor function. The associative subregion receives widespread projections from the prefrontal cortex and serves as a core node in the cognitive control network, regulating cognitive processes such as inhibitory control, set-shifting, and working memory.

High-frequency (>100Hz) deep brain stimulation of the STN (STN-DBS) is a well-established effective treatment for mid-to-late stage PD and can significantly improve motor symptoms. However, long-term high-frequency stimulation may exacerbate cognitive impairment. Recent studies have shown that low-frequency (4-10Hz) STN-DBS can improve cognitive functions such as working memory and verbal fluency in PD patients, but research on its effects in the domain of inhibitory control is lacking. Moreover, different STN subregions are involved in regulating distinct functions, yet previous studies have not differentiated the effects of stimulation targeting specific STN subregions.

Therefore, conducting in-depth research on the effects of different stimulation frequencies applied to distinct STN subregions on inhibitory control function in PD patients is of great significance for exploring ways to improve cognitive impairment in PD and enhance the clinical individualized therapeutic effects of STN-DBS. This study plans to perform high- and low-frequency electrical stimulation of different STN subregions in PD patients who have undergone routine bilateral STN-DBS surgery, collect behavioral indicators during inhibitory control tasks (Arrow Flanker and Stop-Signal) under different stimulation conditions, and through comparative analysis, identify the specific stimulation sites and frequencies that can effectively improve inhibitory control function in PD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80 years old;
2. Diagnosed with idiopathic Parkinson's disease;
3. Meeting the indications for DBS surgery.

Exclusion Criteria:

1. Patient declined to participate in the study;
2. Presence of significant post-DBS complications (e.g., intracranial hemorrhage, cerebral edema, electrode misplacement);
3. Significant psychiatric disorders or dementia (MMSE score <20 for uneducated; <23 for 1-6 years education; <27 for ≥7 years education);
4. Visual or auditory impairment affecting cognitive task performance
5. History of conditions potentially impairing cognitive function.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Behavioral paradigm results | Outcome measures were assessed starting at 5 minutes after each stimulation condition
  1. Arrow Flanker Task : Reaction time for congruent and incongruent trials.

SECONDARY OUTCOMES:
Behavioral paradigm results | Outcome measures were assessed starting at 5 minutes after each stimulation condition
  Stop-Signal Task: Stop-signal reaction time (SSRT).
Motor score | Outcome measures were assessed starting at 5 minutes after each stimulation condition
  MDS-UPDRS III score: The Movement Disorder Society-sponsored Unified Parkinson's Disease Rating Scale Part III (MDS-UPDRS III) is a standardized clinical assessment tool for evaluating motor symptoms in Parkinson's disease (PD). The total score ranges from 0 to 132, with higher scores indicating more severe motor dysfunction, including increased rigidity, bradykinesia (slowed movement), tremor, and postural instability. Conversely, lower scores reflect milder or absent motor impairments, suggesting better motor function and symptom control.

CONTACTS AND LOCATIONS:
Overall Officials: Jianguo Zhang, M.D., Ph.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No